CLINICAL TRIAL: NCT01803243
Title: The Measurement of Spine Dynamics During Gait for the Quantification of Intervention Outcomes in Patients With Different Pathologies
Brief Title: Spine Biomechanics During Gait Following Lower Extremity Treatment in Different Patient Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital Basel (Other)
Collaborators: Swiss Federal Institute of Technology (Other); Bern University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Prof. Reinald Brunner, MD, Doctor in Charge, Neuro-Orthopedics, University Children's Hospital Basel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKBB-Spine-1315-2
Record Dates: First submitted 2013-02-26; First posted 2013-03-04 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Leg Length Inequality; Cerebral Palsy
MeSH Terms: conditions — Leg Length Inequality; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Leg length correction (Experimental): The shorter leg in a sample of 15 patients with structural leg length inequality will be corrected by either a shoe insole or a modified shoe with sole lift.
  Interventions: Other: Shoe insole; Other: Modified shoe with sole lift
- Control of foot position 1 (Experimental): The foot position in in a sample of 15 patients with hemiplegic cerebral palsy will be controlled by an ankle foot orthosis.
  Interventions: Other: Ankle foot orthosis
- Control of foot position 2 (Experimental): The foot position in in a sample of 15 patients with diplegic cerebral palsy will be controlled by an ankle foot orthosis.
  Interventions: Other: Ankle foot orthosis
- Control (No Intervention): A sample of 15 healthy controls from a simultaneously conducted study (UKBB-Spine-1315-1) will be used for comparative purposes.

INTERVENTIONS:
Other: Ankle foot orthosis — Ankle foot orthoses are a common treatment method to control the foot position during walking and to prevent ankle plantar flexion contractures in cerebral palsy patients.
  Arms: Control of foot position 1; Control of foot position 2
Other: Shoe insole — The heel of the shorter leg of the patient is lifted by a shoe insole. This procedure is commonly applied with leg length differences of up to 20mm.
  Arms: Leg length correction
Other: Modified shoe with sole lift — The heel of the shorter leg of the patient is lifted by building up the sole of the shoe (shoe sole lift). This procedure is commonly applied with leg length differences of 20mm and more.
  Arms: Leg length correction

SUMMARY:
Measuring spine dynamics is a necessity in order to better understand gait deviations throughout the whole body and to evaluate treatment effects on spinal movement during gait. However, the full body marker sets that are typically used in opto-electronic 3D gait analyses either disregard the spine entirely or regard it as a rigid structure. Therefore, the purpose of this study is to use an enhanced trunk marker set in order to evaluate the biomechanical effects of lower extremity treatments on spine dynamics in patients with different pathologies.

It has been hypothesized that

1. the enhanced trunk marker set is a reliable method for the measurement of spine dynamics during gait in patients with deviations occurring secondary to leg length inequality.
2. the enhanced trunk marker set is a reliable method for the measurement of spine dynamics during gait in patients that present both primary and secondary deviations such as seen in hemiplegic and diplegic cerebral palsy.
3. treatment by means of either a shoe insole or a modified shoe with sole lift on the shorter side has an effect on spine dynamics during gait in patients with leg length inequality.
4. treatment by means of an ankle foot orthosis to control the foot position has an effect on spine dynamics during gait in patients with hemiplegic and diplegic cerebral palsy.

To verify the hypotheses, instrumented gait analyses with a standard full body marker set and the enhanced trunk marker set will be carried out before and immediately after an orthotic lower extremity treatment in the respective patient group.

ELIGIBILITY:
Leg length inequality patients:

Inclusion Criteria:

* Diagnosed structural leg length inequality (minimum 1% of body height)
* Several different aetiologies (except neurological)
* Able to walk a distance of minimum 50 meters without any assistive device

Exclusion Criteria:

* Leg length inequality due to neurological aetiology
* Structural deformities of the spine
* Obesity (> 95th BMI-per-age percentile)
* Injuries of the locomotor system which led to persistent deformities

Hemiplegic cerebral palsy patients:

Inclusion Criteria:

* Diagnosed hemiplegic cerebral palsy (Gross Motor Function Classification System for Cerebral Palsy (GMFCS): Levels I and II)
* Able to walk a distance of minimum 50 meters barefoot and without any assistive device

Exclusion Criteria:

* Structural deformities of the spine
* Any previous surgical and casting treatments as well as botulinumtoxin treatments within preceding 6 months.
* Obesity (> 95th BMI-per-age percentile)
* Injuries of the locomotor system which led to persistent deformities

Diplegic cerebral palsy patients:

Inclusion Criteria:

* Diagnosed diplegic cerebral palsy (Gross Motor Function Classification System for Cerebral Palsy (GMFCS): Levels I and II)
* Able to walk a distance of minimum 50 meters barefoot and without any assistive device

Exclusion Criteria:

* Structural deformities of the spine
* Any previous surgical and casting treatments as well as botulinumtoxin treatments within preceding 6 months.
* Obesity (> 95th BMI-per-age percentile)
* Injuries of the locomotor system which led to persistent deformities

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Reliability of the enhanced trunk marker set for the measurement of spinal kinematics in patients with leg length inequality and cerebral palsy during gait. | Data will be collected between April 2013 and June 2015. Each patient will be measured before and immediately after an orthotic treatment (both measurements within 1 hour).
  Parameters include lumbar, thoracic and cervical spine curvature angles in the sagittal and frontal planes and segmental rotation angles in the transverse plane.
Immediate changes in spinal kinematics in patients with leg length inequality and cerebral palsy during gait following an orthotic lower extremity treatment. | Data will be collected between April 2013 and June 2015. Each patient will be measured before and immediately after the orthotic treatment (both measurements within 1 hour).
  Parameters include lumbar, thoracic and cervical spine curvature angles in the sagittal and frontal planes and segmental rotation angles in the transverse plane.

SECONDARY OUTCOMES:
Immediate changes in spatio-temporal gait parameters and kinematics and kinetics of peripheral joints in patients with leg length inequality and cerebral palsy during gait following an orthotic lower extremity treatment. | Data will be collected between April 2013 and June 2015. Each patient will be measured before and immediately after the orthotic treatment (both measurements within 1 hour).
  Parameters include gait speed, cadence and single and double limb support as well as angles, torques and powers of peripheral joints in all three planes.

CONTACTS AND LOCATIONS:
Overall Officials: Reinald Brunner, MD, Principal Investigator — University Children's Hospital Basel; Stefan Schmid, PT, PhD, Study Chair — Swiss Federal Institute of Technology / Bern University of Applied Sciences; Silvio Lorenzetti, PhD, DSc, Study Director — Swiss Federal Institute of Technology; Jacqueline Romkes, PhD, Study Director — University Children's Hospital Basel
Locations (1):
- University Children's Hospital Basel, Basel, Switzerland

REFERENCES:
- [Result] Schmid S, Romkes J, Taylor WR, Lorenzetti S, Brunner R. Orthotic correction of lower limb function during gait does not immediately influence spinal kinematics in spastic hemiplegic cerebral palsy. Gait Posture. 2016 Sep;49:457-462. doi: 10.1016/j.gaitpost.2016.08.013. Epub 2016 Aug 12. PMID 27543740